CLINICAL TRIAL: NCT03879694
Title: A Phase I Study of Safety and Immunogenicity of Survivin Long Peptide Vaccine (SurVaxM) in Patients With Metastatic Neuroendocrine Tumors (NETs)
Brief Title: Survivin Long Peptide Vaccine in Treating Patients With Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: NeuroEndocrine Tumor Research Foundation (NETRF) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 79518; NCI-2019-00827 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 79518 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Atypical Carcinoid Tumor; Lung Typical Carcinoid Tumor; Metastatic Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — incomplete Freund's adjuvant; montanide ISA 51; Octreotide; Acetates; Salts; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (SVN53-67/M57-KLH peptide vaccine, octreotide) (Experimental): Patients receive a SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant SC and sargramostim SC on day 0. Treatment repeats every 2 weeks for up to 4 doses in the absence of disease progression or unacceptable toxicity. Patients also receive octreotide acetate IM on day 0. Cycles of octreotide acetate repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who remain free of tumor progression at 6 months and do not develop any regimen-related toxicity or serious adverse events will be eligible to receive additional doses of the vaccine and sargramostim every 3 months, for up to 1 year from the start of treatment.
  Interventions: Biological: Incomplete Freund's Adjuvant; Drug: Octreotide Acetate; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine

INTERVENTIONS:
Biological: Incomplete Freund's Adjuvant — Given SC
  Other Names: Freund's Incomplete Adjuvant; IFA; ISA-51; Montanide ISA 51; Montanide ISA-51
Drug: Octreotide Acetate — Given IM
  Other Names: D-Phenylalanyl-L-cysteinyl-L-phenylalanyl-D-tryptophyl-L-lysyl-L-threonyl-N-[(1R,2R)-2-hydroxy-1-(hyroxymethyl)propyl]-L-cysteinamide, Cyclic (2->7)-disulfide, Acetate (Salt); Longastatin; Longastatina; Samilstin; Sandostatin; Sandostatin Lar Depot; Sandostatina; Sandostatine; SMS 201-995; SMS 201-995 AC
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: SVN53-67/M57-KLH Peptide Vaccine — Given SC

SUMMARY:
This phase I trial studies the side effects of survivin long peptide vaccine and how it works with the immune system in treating patients with neuroendocrine tumors that have spread to other parts of the body (metastatic). Tumor cells make proteins that are not usually produced by normal cells. The body sees these proteins as not belonging and sends white blood cells called T cells to attack the tumor cells that contain these proteins. By vaccinating with small pieces of these proteins called peptides, the immune system can be made to kill tumor cells. Giving survivin long peptide vaccine to patients who have survivin expression in their tumors may create an immune response in the blood that is directed against neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety, tolerability and toxicity of SVN53-67/M57-KLH peptide vaccine (SurVaxM) in emulsion with incomplete Freund's adjuvant (montanide ISA 51) and given subcutaneously with sargramostim (granulocyte macrophage-colony-stimulating factor [GM-CSF]) in combination with a somatostatin analogue, octreotide acetate (Sandostatin LAR) in patients with survivin positive metastatic neuroendocrine tumors (NETs).

SECONDARY OBJECTIVES:

I. To determine clinical benefit (including complete response, partial response and stable disease as defined by Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) at 6 months, 9 months and 12 months from study entry.

II. To evaluate the immunogenicity of SurVaxM in NETs by measuring anti-survivin antibody levels and anti-tumor T-cell responses in peripheral blood.

III. To determine time to progression (TTP) compared to prior to study entry, in patients with metastatic NETs treated with SurVaxM.

EXPLORATORY OBJECTIVES:

I. To explore immune markers associated with clinical responses to SurVaxM in peripheral blood of NETs patients.

OUTLINE:

Patients receive a SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant subcutaneously (SC) and sargramostim SC on day 0. Treatment repeats every 2 weeks for up to 4 doses in the absence of disease progression or unacceptable toxicity. Patients also receive octreotide acetate intramuscularly (IM) on day 0. Cycles of octreotide acetate repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who remain free of tumor progression at 6 months and do not develop any regimen-related toxicity or serious adverse events will be eligible to receive additional doses of the vaccine and sargramostim every 3 months, for up to 1 year from the start of treatment.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a Karnofsky performance status >= 70 or Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (i.e. the patient must be able to care for himself/ herself with occasional help from others).
* Pathologically confirmed diagnosis of neuroendocrine tumor of gastrointestinal, pancreatic or lung origin.
* Patients who have been on somatostatin analogues (SSA) may continue to take SSA while on study treatment.
* Patients must have documented progression within the last six months on CT or MRI scans performed at least four weeks apart per RECIST v1.1 criteria. In the case of retreatment, progression may be defined by the treating provider (e.g., clinical, radiographic, biochemical).
* Archival neuroendocrine tumor tissue must test positive for survivin presence by clinical immunohistochemistry prior to study enrollment
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained within 14 days prior to enrollment).
* Platelets >= 100 x 10^9/L (obtained within 14 days prior to enrollment).
* Hemoglobin (Hgb) > 9g/dL (obtained within 14 days prior to enrollment).
* Plasma total bilirubin: =< 1.5 x upper limit of normal (ULN) (obtained within 14 days prior to enrollment).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 4 x ULN (obtained within 14 days prior to enrollment).
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices, which carries a significant risk of bleeding in investigator's opinion).
* Creatinine =< 1.8 mg/dL (obtained within 14 days of enrollment).
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and, have a negative pregnancy test prior to starting study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* The patient must not have received any immunotherapy for any malignancy,as long as it was > 3 months prior to study start.
* Patients with serious concurrent infection or medical illness, which in the treating physicians' opinion would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Patients who are pregnant or breast-feeding.
* Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for at least 3 years are eligible for this study.
* Known history of an autoimmune disorder.
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness.
* Previous local therapy (e.g. chemo-embolization, bland, or radio-embolization) is allowed if completed > 6 weeks prior to randomization. For subjects who received local therapy prior to randomization, there must be documented growth of measurable disease within the embolization field prior to study.
* Unwilling or unable to follow protocol requirements.
* Systemic corticosteroid therapy > 2 mg of dexamethasone or equivalent per day at study entry.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.
* Received an investigational agent within 30 days prior to enrollment.
* Clinically significant cardiac arrhythmia, bradycardia, tachycardia that would compromise patient safety or the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of SVN53-67/M57-KLH peptide vaccine in combination with octreotide acetate in patients with neuroendocrine tumors | Up to 15 months
  Will be assessed with National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will consider a toxicity to be an adverse event that is possibly, probably or definitely related to treatment. The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. Will be quantified using the observed rates of the adverse events, serious adverse events (SAE) and regimen limiting toxicities. Toxicity rates will be described using upper 1-sided 95% Jeffreys binomial confidence intervals.

SECONDARY OUTCOMES:
Immunogenicity of SVN53-67/M57-KLH peptide vaccine | Baseline up to 15 months
  Survivin-specific CD8+ responses will be measured individually at baseline, 12 weeks and end of-study. These measures will be summarized by descriptive statistics (means, medians, quartiles, etc.). Confidence intervals will be constructed for the median and the mean. Exploratory graphical analysis will be used to discover associations among variables.
Immunogenicity of SVN53-67/M57-KLH peptide vaccine | Baseline up to 15 months
  Anti-survivin antibody (humoral) responses will be measured individually at baseline, 12 weeks and end of-study. These measures will be summarized by descriptive statistics (means, medians, quartiles, etc.). Confidence intervals will be constructed for the median and the mean. Exploratory graphical analysis will be used to discover associations among variables.
Rate of progression | Up to 15 months
  Will be based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 on computed tomography scan and comparison rate prior to start of treatment.
Clinical benefit | Up to 12 months
  Will be assessed with RECIST v1.1. Clinical Benefit (CB) is defined as number of patients having best overall response as complete response (CR), partial response (PR) or stable disease (SD). The estimated distribution of CB will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available.
Time to progression (TTP) | From enrollment to first documented progression per RECISTv1.1, assessed up to 15 months
  The TTP of each patient will be compared to TTP prior to study entry. The analysis will be descriptive and reported separately for each patient.
Overall response rate (ORR) | Up to 15 months
  Measured by RECIST v1.1.
Duration of response (DOR) | Up to 15 months
  Measured by RECIST v1.1.

OTHER OUTCOMES:
Serum levels of chromogranin A, serotonin and 5-HIAA | Baseline up to 15 months
  Exploratory graphical analysis will be used to discover associations among variables.
Serum levels of serotonin and 5-HIAA | Baseline up to 15 months
  Exploratory graphical analysis will be used to discover associations among variables
Serum levels of 5-HIAA | Baseline up to 15 months
  Exploratory graphical analysis will be used to discover associations among variables

CONTACTS AND LOCATIONS:
Overall Officials: Jasmeet Kaur, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States